CLINICAL TRIAL: NCT07305844
Title: Open-label, Single-arm Study to Assess the Colonization Kinetics of Clinician- Administered Vaginal Live Biotherapeutic Product Containing Multiple Strains of Lactobacillus Crispatus.
Brief Title: Impact of Clinician-administered Vaginal Live Biotherapeutic Product
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Caroline Mitchell (Other)
Responsible Party: Sponsor-Investigator, Caroline Mitchell, Associate Professor, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMRC-002
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Re-challenge (Experimental): Administration of LC106 in clinic, for three days
  Interventions: Drug: LC106

INTERVENTIONS:
Drug: LC106 — This is a 6-strain L. crispatus vaginal live biotherapeutic tablet

SUMMARY:
This is an open-label, single-arm, Phase Ib trial assessing the consistency of response and colonization kinetics of a vaginally inserted live biotherapeutic intervention with optimized adherence.

DETAILED DESCRIPTION:
In this study investigators will enroll participants from the VIBRANT study who received active study product and test the vaginal microbiome. If a participant does not have a Lactobacillus predominant vaginal microbiome, they will re-dose with LC106 in the clinic for three days in a row. This will allow understanding of how consistent the response to LC106 is, and whether directly monitored administration improves results.

ELIGIBILITY:
Inclusion Criteria:

* Previous participant in the VIBRANT study, randomized to active LBP
* Nugent score 4-10

Exclusion Criteria:

* Infection requiring antibiotics detected on screening labs
* Use of oral or vaginal antibiotics in the 30 days prior to screening
* Use of an oral or vaginal probiotic in the 30 days prior to screening

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Rate of colonization with LBP isolates | 5 weeks
  Detection of at least one isolate from the LBP with at least 5% relative abundance by metagenomics, or a combination of isolates at 10% or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Mitchell, MD, MPH, Principal Investigator — Massachusetts General Hospital; Disebo Potloane, MD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- CAPRISA, Vulindlela, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Microbial sequences
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At the time of publication of study results
Access Criteria: THe microbial reads will be posted on a public site, such as the Short Read Archive